CLINICAL TRIAL: NCT02805608
Title: Phase II Trial: uPAR PET/CT and FDG PET/MRI for Preoperative Staging of Bladder Cancer
Brief Title: uPAR PET/CT and FDG PET/MRI for Preoperative Staging of Bladder Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Dorthe Skovgaard, MD, Phd, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AK2016-1
Record Dates: First submitted 2016-06-13; First posted 2016-06-20 (Estimated); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- uPAR PET/CT and FDG PET/MR (Experimental): One injection of 68Ga-NOTA-AE105 followed by PET/CT and on a separate day one injection of 18F-FDG followed by PET/MRI. Both scans will be evaluated for possible regional lymph node metastases.
  Interventions: Drug: Injection of 68Ga-NOTA-AE105; Drug: Injection of 18F-FDG; Device: Positron Emission Tomography and CT; Device: Positron Emission Tomography and MRI

INTERVENTIONS:
Drug: Injection of 68Ga-NOTA-AE105 — One injection intravenously of 68Ga-NOTA-AE105
Drug: Injection of 18F-FDG — One injection intravenously of 18F-FDG
Device: Positron Emission Tomography and CT — Following of injection of 68Ga-NOTA-AE105 the patients will be PET/CT scanned starting 20 minutes post injection
Device: Positron Emission Tomography and MRI — Following injection of 18F-FDG the patients will be PET/MRI scanned starting 60 minutes post injection

SUMMARY:
The sensitivity and specificity of uPAR PET/CT with the radioligand 68GaNOTA-AE105 and FDG PET/MRI for preoperative detection of regional lymph node metastases in urinary bladder cancer

DETAILED DESCRIPTION:
The sensitivity and specificity of 68Ga-NOTA-AE105 PET/CT and FDG PET/MRI for detection of regional lymph node metastases will be tested by observer-blinded readings and compared to diagnostic performance of conventional preoperative procedure. The reference test will be histopathology of lymph nodes obtained by operative lymph node dissection based on 6 regions. The suspected lymph nodes will be assigned to 6 regions based on the images. During the following operation the lymph nodes will be removed and analysed in each of these regions.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-verified urinary bladder cancer
* The participants must be capable of understanding and giving full informed written consent age above 18 years

Exclusion Criteria:

* Pregnancy
* Lactation/breast feeding
* Age above 85 years old
* Weight above 140 kg
* Treatment with neoadjuvant chemotherapy
* Known allergy towards 68Ga-NOTA-AE105
* Other malignant disease within last 5 years, except for non-melanoma

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
uPAR PET/CT: regional lymph node metastases | evaluated on uPAR-PET/CT scan performed within 1 hour following injection of 68Ga-NOTA-AE105
  Sensitivity of uPAR-PET/CT detection of regional lymph node metastases by 68Ga-NOTA-AE105 PET/CT
FDG PET/MRI: regional lymph node metastases | evaluated on FDG PET/MRI performed within 1 hour following injection of 18F-FDG
  Sensitivity of FDG-PET/MRI for detection of regional lymph node metastases

SECONDARY OUTCOMES:
uPAR PET/CT: Number of lymph node metastases | evaluated on uPAR-PET/CT performed within 1 hour following injection of 68Ga-NOTA-AE105
  Number of true positive lymph node metastases detected by uPAR-PET/CT
FDG PET/MRI: Number of lymph node metastases | evaluated on FDG PET/MRI performed within 1 hour following injection of 18F-FDG
  Number of true positive lymph node metastases detected by FDG-PET/MRI
uPAR PET/CT: sensitivity for detection of distant metastases | evaluated on uPAR-PET/CT performed within 1 hour following injection of 68Ga-NOTA-AE105
  Sensitivity for detection of true positive distant metastases by uPAR-PET/CT
FDG PET/MRI: sensitivity for detection of distant metastases | evaluated on uPAR-PET/CT performed within 1 hour following injection of 18F-FDG
  Sensitivity for detection of true positive distant metastases by FDG-PET/MRI

CONTACTS AND LOCATIONS:
Overall Officials: Dorthe Skovgaard, Md, PhD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Department of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No